CLINICAL TRIAL: NCT01206166
Title: A Randomized Trial of Supplemental Parenteral Nutrition in Under and Over Weight Critically Ill Patients: The TOP UP Trial (Pilot)
Brief Title: Trial of Supplemental Parenteral Nutrition in Under and Over Weight Critically Ill Patients (TOP-UP)
Acronym: TOP-UP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment rates.
Sponsor: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Daren K. Heyland, Director, Clinical Evaluation Research Unit at Kingston General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TOP-UP
Record Dates: First submitted 2010-09-14; First posted 2010-09-21 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Critical Illness; Acute Respiratory Failure
Keywords: Randomized trial; Parental nutrition; Enteral nutrition; Intensive care unit; BMI < 25 or ≥ 35
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enteral Nutrition + Parenteral Nutrition (Experimental): Enteral nutrition with the addition of parenteral supplementation (Olimel 5.7%E/N9E).
  Interventions: Drug: Olimel (5.7%E / N9E)
- Enteral Nutrition Only (No Intervention): Enteral nutrition only - no intervention

INTERVENTIONS:
Drug: Olimel (5.7%E / N9E) — OLIMEL(Amino Acids, Dextrose, Lipids, with / without Electrolytes) is indicated for parenteral nutrition for adults when oral or enteral nutrition is impossible, insufficient or contraindicated.
  Other Names: Olimel
  Arms: Enteral Nutrition + Parenteral Nutrition

SUMMARY:
The specific aim of the proposed study is to conduct a pilot study involving 160 critically-ill lean and obese patients enrolled at 11 sites in Canada, the United States of America, Belgium and France in order to:

Specific Aims

* Confirm that we can achieve a clinically significant difference in calorie and protein intake between the two intervention groups.
* Estimate recruitment rate i.e. number of eligible and enrolled patients per month per site.
* Evaluate the safety, tolerance, and logistics around providing supplemental PN in the study population in the context of a multicenter trial, e.g.

  * To ensure adequate glycemic control in both groups.
  * To ensure that the other metabolic consequences of the feeding strategies are minimized.
  * To establish adequate compliance with study protocols and completion of case report forms

A secondary aim of this pilot study will be:

• To explore the effect of differential effects of calorie and protein delivery on muscle and mass function.

DETAILED DESCRIPTION:
Background

Critically ill patients are often hypermetabolic and can rapidly become nutritionally compromised. Malnutrition is prevalent in these patients and has been associated with increased morbidity and mortality. Standard nutrition therapy, i.e. provision of calories, protein and other nutrients consists primarily of enteral nutrition (via a feeding tube into the gastrointestinal tract), parenteral nutrition (via an intravenous tube into the blood), or occasionally a combination of both.

However, the provision of nutrition is sub-optimal and the majority of critically-ill patients do not meet nutritional requirements. Recent studies report that average energy intakes of critically ill patients are only 49% to 70% of calculated requirements. Despite repeated, sustained efforts over the past few years, the investigators have not significantly improved the amount of calories delivered via the enteral route. This leads us to conclude that if the investigators are to be successful at increasing the provision of calories and protein to patients at-risk, the investigators will have to supplement the calories via the parenteral route.

Critically ill patients that are at extremes of weight are at a higher nutritional risk and have higher mortality rates. A recent International multicenter observational study of 2772 ICU patients from 165 ICUs showed a significant inverse linear relationship between the odds of mortality and total daily calories received. Increased amounts of calories was most important for the BMI < 20 group followed by the BMI 20 -< 25 group and BMI > 35 group with no benefit of increased calorie intake for patients in the BMI 25 -< 35 group. Feeding an additional 1000 kcals almost halved the odds of 60-day mortality in patients with a BMI < 25 or > 35. Similar results were observed for feeding an additional 30 grams of protein per day.

Thus, a prospective randomized trial is warranted to confirm our hypothesis that in patients with a BMI of < 25 and those with a BMI > 35 increasing the provision of more energy and protein can impact clinical outcomes. The results of this study will serve to answer some fundamental questions with regards to impact of amount of energy and protein delivered to nutritional at-risk ICU patients and will inform current practice.

Study Intervention:

Patients will be randomized to one of 2 interventions: enteral nutrition alone or enteral nutrition plus parenteral nutrition (supplemental PN group).

ELIGIBILITY:
Inclusion Criteria:

* Critically ill adult patient (≥ 18 years) admitted to ICU
* Has acute respiratory failure (ARF) i.e. expected to remain mechanically ventilated for more than 48 hours
* Expected ICU dependency of 5 or more days
* On or expected to initiate enteral nutrition within 7 days of ICU admission
* BMI <25 or ≥ 35 based on pre-ICU actual or estimated dry weight

Exclusion Criteria:

* >72 hours from admission to ICU to time of consent
* Not expected to survive an additional 48 hrs from screening evaluation
* A lack of commitment to full aggressive care (anticipated withholding or withdrawing treatments in the first week but isolated DNR acceptable)
* Patients already receiving PN at screening
* Absence of All gastrointestinal risk factors, defined as:

  1. High Apache II Score (>20)
  2. On more than 1 vasopressor or increasing doses or vasopressors
  3. Receiving continuous infusion of narcotics
  4. High nasogastric/orogastric output (>500 mL over 24 hours)
  5. Recent surgery involving esophagus, stomach, or small bowel OR peritoneal contamination with bowel contents
  6. Pancreatitis
  7. Multiple gastrointestinal investigations
  8. Recent history of diarrhea/C. Difficile
  9. Surgical patients with future surgeries planned
  10. Ruptured or dissected abdominal aortic aneurysm
* Patients admitted with diabetic ketoacidosis or non-ketotic hyperosmolar coma
* Pregnant or lactating patients
* Patients with clinical fulminant hepatic failure
* Patients with Cirrhosis Child's Class C Liver Disease (except those on a transplant list or transplantable)
* Dedicated port of central line not available
* Known allergy to study nutrients (soy, eggs or olive products)
* Enrolment in another industry sponsored ICU intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-06; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daren K. Heyland, MD, Study Chair — Clinical Evaluation Research Unit, Kingston General Hospital
Locations (12):
- United States (7):
  - University of Colorado DHSC, Boulder, Colorado
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio
  - The Ohio State Univsersity Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Texas Health Science Center, Houston, Texas
- Erasme University Hospital, Brussels, Belgium
- Canada (3):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta
- Nouvel Hôpital Civil, Strasbourg, France

REFERENCES:
- [Background] Alberda C, Gramlich L, Jones N, Jeejeebhoy K, Day AG, Dhaliwal R, Heyland DK. The relationship between nutritional intake and clinical outcomes in critically ill patients: results of an international multicenter observational study. Intensive Care Med. 2009 Oct;35(10):1728-37. doi: 10.1007/s00134-009-1567-4. Epub 2009 Jul 2. PMID 19572118
- [Background] Villet S, Chiolero RL, Bollmann MD, Revelly JP, Cayeux R N MC, Delarue J, Berger MM. Negative impact of hypocaloric feeding and energy balance on clinical outcome in ICU patients. Clin Nutr. 2005 Aug;24(4):502-9. doi: 10.1016/j.clnu.2005.03.006. PMID 15899538
- [Background] Krishnan JA, Parce PB, Martinez A, Diette GB, Brower RG. Caloric intake in medical ICU patients: consistency of care with guidelines and relationship to clinical outcomes. Chest. 2003 Jul;124(1):297-305. doi: 10.1378/chest.124.1.297. PMID 12853537
- [Background] Hise ME, Halterman K, Gajewski BJ, Parkhurst M, Moncure M, Brown JC. Feeding practices of severely ill intensive care unit patients: an evaluation of energy sources and clinical outcomes. J Am Diet Assoc. 2007 Mar;107(3):458-65. doi: 10.1016/j.jada.2006.12.012. PMID 17324665
- [Background] Dhaliwal R, Jurewitsch B, Harrietha D, Heyland DK. Combination enteral and parenteral nutrition in critically ill patients: harmful or beneficial? A systematic review of the evidence. Intensive Care Med. 2004 Aug;30(8):1666-71. doi: 10.1007/s00134-004-2345-y. Epub 2004 Jun 8. PMID 15185069
- [Derived] Wischmeyer PE, Hasselmann M, Kummerlen C, Kozar R, Kutsogiannis DJ, Karvellas CJ, Besecker B, Evans DK, Preiser JC, Gramlich L, Jeejeebhoy K, Dhaliwal R, Jiang X, Day AG, Heyland DK. A randomized trial of supplemental parenteral nutrition in underweight and overweight critically ill patients: the TOP-UP pilot trial. Crit Care. 2017 Jun 9;21(1):142. doi: 10.1186/s13054-017-1736-8. PMID 28599676

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enteral Nutrition + Parenteral Nutrition | Enteral Nutrition Only
Started | 73 | 52
Completed | 71 | 49
Not Completed | 2 | 3
Not completed — No evaluable data | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enteral Nutrition + Parenteral Nutrition | Enteral Nutrition Only | Total
Number analyzed (Participants) | 73 | 52 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (16.2) | 55.8 (19.8) | 55.45 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 31 | 65
  Male | 39 | 21 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 65 | 46 | 111
  Black or African American | 4 | 2 | 6
  Native Hawaiian or Pacific Islander | 2 | 0 | 2
  Native | 2 | 0 | 2
  unknown/unreported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Calorie & Protein Intake 7 Days Post Randomization
Description: Amount of calories & protein received as a percentage of prescribed.
Time Frame: 7 days post randomization
Population: ICU patients
Measure: Mean (Standard Deviation); unit: percentage of prescribed
Groups:
- EN Only: Enteral nutrition no intervention
Arm/Group | EN Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 71 | 49
percentage of prescribed
  calories in first 7 days | 69 (28) | 95 (13)
  protein in first 7 days | 64 (26) | 86 (16)

2. Secondary Outcome: 6 Month Mortality
Description: Kaplan-Meier estimate.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Groups:
- Enteral Nutrition Only: Enteral nutrition no intervention
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
percentage of participants | 27.5 | 29.5

3. Secondary Outcome: ICU Mortality
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
Participants | 13 | 7

4. Secondary Outcome: Hospital Mortality
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
Participants | 17 | 8

5. Secondary Outcome: Duration of ICU Stay
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
days | 12.6 [8.1 to 18.7] | 12.8 [7.9 to 17.8]

6. Secondary Outcome: Duration of Hospital Stay
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
days | 24 [16.6 to 38.9] | 23.5 [17.5 to 34.7]

7. Secondary Outcome: Duration of Mechanical Ventilation
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
days | 8.3 [3.8 to 13.3] | 6.5 [3.9 to 14.1]

8. Secondary Outcome: Development of ICU-acquired Infections
Time Frame: ICU discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
Participants | 23 | 14

9. Secondary Outcome: SF36-Physical Functioning Domain
Description: The SF-36 physical function domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Enteral Nutrition Only: Enteral Nutrition only-no intervention
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 39.4 (34.3) | 34.8 (31.5)

10. Secondary Outcome: SF-36 Physical Functioning Domain
Description: The SF-36 physical function domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 39.3 (34) | 50.8 (36.5)

11. Secondary Outcome: Functional Status at Hospital Discharge
Time Frame: hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
Participants
  hand grip: Pt died | 17 | 8
  hand grip: Unable to do | 12 | 5
  hand grip: Refused to do | 3 | 3
  hand grip: Done | 22 | 17
  hand grip: Missed | 16 | 12
  hand grip: Unknown reason | 1 | 4
  hand grip: use ICU | 2 | 3
  6min walk test: Pt died | 17 | 8
  6min walk test: Unable to do | 31 | 20
  6min walk test: Refused to do | 3 | 3
  6min walk test: Done | 9 | 9
  6min walk test: Missed | 12 | 9
  6min walk test: Unknown reason | 1 | 3
  6min walk test: use ICU | 0 | 0

12. Primary Outcome: Calorie & Protein Intake in First 27 Days
Description: Amount of calories & protein received as a percentage of prescribed.
Time Frame: first 27 days
Population: ICU patients
Measure: Mean (Standard Deviation); unit: percentage of prescribed
Arm/Group | EN Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 71 | 49
percentage of prescribed
  calories in first 27 days | 72 (25) | 90 (16)
  protein in first 27 days | 68 (25) | 82 (19)

13. Secondary Outcome: SF36 Role Physical Domain
Description: The SF-36 role physical function domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 30.2 (31.8) | 32.8 (32.6)

14. Secondary Outcome: SF36 Pain Index Domain
Description: The SF-36 pain index domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 59.1 (28.8) | 66.4 (27.3)

15. Secondary Outcome: SF36 General Health Perceptions Domain
Description: The SF-36 general health perceptions domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 61.2 (18.3) | 49.5 (24.3)

16. Secondary Outcome: SF36 Vitality Domain
Description: The SF-36 vitality domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 52.8 (21.4) | 51 (21.7)

17. Secondary Outcome: SF36 Social Functioning Domain
Description: The SF-36 social functioning domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 60.4 (31.8) | 56.5 (28.2)

18. Secondary Outcome: SF36 Role-emotional Domain
Description: The SF-36 role-emotion domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 63.2 (34.6) | 65.3 (34.4)

19. Secondary Outcome: SF36 Mental Health Index Domain
Description: The SF-36 mental health index domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 72.9 (18.7) | 76.1 (18.5)

20. Secondary Outcome: SF36 Standardized Physical Component Scale
Description: The SF36 Standardized Physical Component Scale has been scaled to have a mean of zero and standard deviation of 10 in a general US population. Higher scores indicate better HRQoL.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 35.3 (10.8) | 33.3 (10.1)

21. Secondary Outcome: SF36 Standardized Mental Component Scale
Description: The SF36 Standardized Mental Component Scale has been scaled to have a mean of zero and standard deviation of 10 in a general US population. Higher scores indicate better HRQoL.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 50 (10.5) | 51.5 (10)

22. Secondary Outcome: SF-36 Role-physical Domain
Description: The SF-36 mental health index domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 40.2 (33.1) | 47.5 (33.4)

23. Secondary Outcome: SF-36 Pain Index Domain
Description: The SF-36 mental health index domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 52.5 (31) | 68.6 (28.2)

24. Secondary Outcome: SF-36 General Health Perceptions Domain
Description: The SF-36 general health perceptions domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 50.9 (20.6) | 56.8 (26.2)

25. Secondary Outcome: SF-36 Vitality Domain
Description: The SF-36 vitality domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 47.8 (21.2) | 59.1 (21.7)

26. Secondary Outcome: SF-36 Social Functioning Domain
Description: The SF-36 social functioning domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 50.4 (32.2) | 68.8 (32.6)

27. Secondary Outcome: SF-36 Role-emotional Domain
Description: The SF-36 role-emotional domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 52.2 (41) | 72.1 (30.3)

28. Secondary Outcome: SF-36 Mental Health Index Domain
Description: The SF-36 mental health index domain ranges from 0-100. Higher scores indicate better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 66.1 (22.5) | 70.5 (24.9)

29. Secondary Outcome: SF-36 Standardized Physical Component Scale
Description: as for outcome 20
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 35.8 (11.2) | 39.3 (10.2)

30. Secondary Outcome: SF-36 Standardized Mental Component Scale
Description: as for outcome 21
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteral Nutrition Only | Enteral Nutrition + Parenteral Nutrition
Number analyzed (Participants) | 73 | 52
score on a scale | 43.2 (14.8) | 49 (13.5)

ADVERSE EVENTS:
Time Frame: 28 days
Description: Given the acuity of illness of critically ill patients, adverse events (defined as any untoward medical occurrences in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment) will not be collected.
Arm/Group | Enteral Nutrition + Parenteral Nutrition | Enteral Nutrition Only
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
due to slower than anticipated enrollment and the upcoming end of the funding from the National Institutes of Health the study was prematurely terminated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No